CLINICAL TRIAL: NCT02186327
Title: Community Coaching: Integrative Health Coaching Initiative for Behavior Change and Assessment of Perceived Needs in the Community Setting
Brief Title: Integrative Health Coaching in Community Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Pro00054909
Record Dates: First submitted 2014-07-02; First posted 2014-07-10 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-01

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: Integrative Health Coaching
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): The control arm will continue to receive standard care as they did prior to enrollment.
- Integrative health coaching (Experimental): Subjects in this arm will receive 6 sessions of integrative health coaching over a 3 month period, in addition to standard care.
  Interventions: Behavioral: Integrative Health Coaching

INTERVENTIONS:
Behavioral: Integrative Health Coaching — Coaching sessions will guide subjects in establishing and maintaining behavior change goals related to their health and overall well-being.
  Arms: Integrative health coaching

SUMMARY:
This study examines a pilot project to introduce integrative health coaching to two community clinical sites, Healing with CAARE Inc. and the Healthy Lifestyles program at Duke Pediatrics. 10 participants and 10 controls will be referred for enrollment at each site (n=20 per site) by on-site personnel, and 6 coaching sessions will be provided over a 3-month period at no cost by coaching trainees completing their certification hours. Pre and post measurements of BMI, patient activation, and perceived interpersonal support will be collected and analyzed for interaction effects. Qualitative process evaluation will be conducted as a thematic analysis via guided interviews with stakeholders and participants, using the "RE-AIM" framework. Feasibility measures will include recruitment of both coaches and clients, subject/client retention, and number and duration of coaching sessions completed. Finally, a subset of the CAARE Inc. cohort will be consented to participate in a post-intervention focus group that addresses the impact of coaching on perception of health-related resources and needs in the community.

Primary Hypotheses:

Integrative health coaching will be a feasible intervention in both community and clinical settings, in terms of required resources, patient or client adherence, and satisfaction by community stakeholders, including providers and participants.

Additional hypotheses:

Individuals who receive integrative health coaching sessions as an adjunct to their standard medical care will see improvements in patient activation and perception of interpersonal supports, when compared to controls.

Individuals who receive integrative health coaching (or in the case of the pediatric cohort, children of individuals who receive coaching) will see minor improvements in BMI over the study period when compared to controls.

DETAILED DESCRIPTION:
Integrative health coaching, based on a curriculum designed and implemented by Duke Integrative Medicine, uses a patient-centered approach that features elements of accountability, self-discovery, and patient-driven goals. It strives to empower patients to enact lifestyle changes situated in the context of their lives, and invites them to identify intrinsic values that might help guide those choices This type of approach is rooted in validated theories of health psychology. Preliminary work using IHC has found this new approach to be effective for improving lifestyle behaviors (diet, exercise, medication adherence) with concomitant improvements in glycemic control in type 2 diabetes, and for reducing the risk of cardiovascular disease (CVD) in patients with traditional risk factors. In addition, program outcomes suggest reduced healthcare spending in patients enrolled in IHC. A large trial to evaluate how this approach will perform in the primary care setting is currently ongoing.

Health coaching and health literacy efforts that are "community-based" or take place in community settings have also been evaluated for effectiveness as well as feasibility and acceptability. Approaches utilized include telephonic coaching and peer coaches, often in an effort to provide increased accessibility. These studies highlight diverse coaching interventions with mixed results. There are no studies of Integrative Health Coaching implemented in non-profit community settings.

Study Procedures

Baseline visit - After screening to confirm eligibility, an in-person baseline visit will be organized with the participant, during which full consent will be obtained. Following subject consent, each participant will be asked to fill out a brief survey instrument on paper consisting of the ISEL-12 and PAM (or Parent PAM for the Healthy Lifestyles cohort). Participants (in the case of the Healthy Lifestyles cohort, pediatric participants and not parents or guardians) will then be weighed without shoes or outer garments using a zeroed electronic scale. Weight will be recorded to the nearest tenth of a pound. Height will be recorded to the nearest tenth of a centimeter using a stadiometer. Body mass index (BMI) will be calculated from these measurements using the conversion formula BMI = weight (kg)/ height (m2). Randomization will occur after collecting baseline measures. If randomized to receive health coaching, the participant (or parent) will receive a handout briefly describing what to expect from their health coaching sessions and how to best prepare. They will also be asked to fill out a "Current and Desired States" form, which is part of the IHC coaching model and will be passed along to coaches for use in the first session.

Integrative Health Coaching Sessions - After completing the baseline visit, each participant randomized to coaching will be scheduled for an initial telephone call (~ 60-75 minutes in length) to discuss the role of a health coach, when and how s/he may be contacted by participants, and an initial participant self-assessment of health perceptions and goals. This self-assessment creates the foundation for the personalization of the behavioral intervention. From this point, participants will schedule weekly to biweekly (~ 30-45 minute) calls with their health coach, for a total of 6 coaching calls over a 3-month intervention period. For the Healthy Lifestyles cohort, all telephonic coaching sessions and activities conducted therein will be directed towards the parent or guardian providing consent. While family health goals and the child's weight management may be anticipated areas of focus in these sessions, coaches and clients will not be limited to any particular topics of discussion.

Participants may initiate coaching sessions from their own personal phone, or by using a landline extension on site at CAARE Inc. or Healthy Lifestyles during business hours, depending on which is more convenient for their schedule and budget. This protocol provides no reimbursement for inadvertent phone charges.

Post-intervention follow-up meeting - Three months following baseline (+ or - one week) and after 6 coaching sessions for the IHC group, participants will meet with a member of the research team to complete the same survey instruments from the baseline visit, and to reassess height and weight, using identical methods to those at baseline. At this time, participants randomized to the IHC group will also have the opportunity to offer recorded feedback regarding their experience in a coaching intervention. This feedback will be solicited via an interview guide of pre-drafted questions, after which the participant will have the opportunity to add additional comments. At this point, unless the participant is part of the subset allocated to the focus group (see below), his/her role in the study is completed. After the post-intervention survey has been completed, coaches and clients may agree to continue sessions on an individual basis, although coaches-in-training must clearly communicate that further sessions are not part of the study.

Focus Group regarding impact of coaching on community needs assessment - This portion of the study will recruit a subset of those participants enrolled from the Healing with CAARE Inc. site. All participants previously enrolled, consented and randomized to receive health coaching will be asked to participate in a focus group session of about 1.5 hours regarding community needs assessment; the target participatory goal is 6-8 participants. The session will take place following post-intervention data collection for all participants who received coaching. It will be guided around a series of questions detailed in a separate document, and centered around data from the 2013 State of the County Health Report and 2013 Community Health Assessment Survey Results conducted and reported by the Durham County Health Department (DCHD) and Partnership for a Healthy Durham. 32 Participants will be invited to comment on the results of these assessments relative to their personal experiences, and to offer their perspectives on community needs, current resources or areas for improvement regarding health and wellness. They will also be asked about their experiences in using community resources or identifying community or environmental barriers through their behavior change efforts while receiving coaching. Participants will be asked whether and how their perspectives on community needs or available resources may have changed following coaching, and if and how they intend to utilize or advocate for community resources in the future.

Post-Intervention Qualitative Evaluation In order to learn as much as possible from this community engagement project, after completion of the study intervention, interviews will be conducted with the coaches that delivered the interventions as well as clinical and administrative staff of the respective community sites. These interviews will take place in small groups or individually and may include briefer, follow-up conversations with the same individuals by phone or in person, to clarify responses as needed. The interviews will be recorded for the purposes of subsequent review and analysis. Participants in the interviews will be identified only by their role in the study in any written analysis of interview content.

The interviews will be structured around a series of interview guides, each of which is composed of a series of questions directed at the health coaches, and community staff or providers who referred patients. Participants will also have an opportunity to draft their own questions regarding the study, and common themes of these questions will be explored further in the group conversation.

Interviews will also be conducted with study participants individually, as outlined above, at the time of their post-intervention follow-up visit. As in the provider and staff interviews, the participant interviews will also be structured around interview guide questions, with an opportunity for participants to draft additional questions or share feedback beyond the question prompts.

The interviews will provide feedback regarding feasibility, delivery, resources utilized, and interprofessional communication throughout the study. Specifically, the areas addressed will include reach, effectiveness, adoption, implementation and maintenance, as have been outlined in previous studies and briefs.

ELIGIBILITY:
Inclusion Criteria:

Site one:

* 18 years or over
* able to speak and understand English
* able and willing to give informed consent

Site two (pediatric):

* pediatric participant is 5-12
* patient is in care of parent or guardian willing to participate in study intervention and complete baseline and post-intervention surveys and interviews
* both pediatric patient and parent/guardian can speak and understand English
* parent/guardian is able and willing to provide consent (pediatric patients age 12 will also provide assent)

Exclusion Criteria:

* inability to ambulate or participate in physical activity
* serious chronic disease related complications or conditions that could significantly affect study outcomes (currently treated cancer, renal failure, CVA with residual effects on functioning)
* concurrent participation in a lifestyle-based intervention study for chronic disease or health behaviors

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Subject attrition rate | 3 months from baseline
  As establishing feasibility is a primary purpose of this study, subject attrition will serve as one primary outcome measure.
Duration (in minutes) of coaching sessions. | 3 months from baseline
  In order to establish subject exposure to the main study intervention and to establish feasibility, number and duration of completed sessions will be measured.
Subject and site personnel process evaluation (reach, effectiveness, adoption, implementation, and maintenance (RE-AIM)) following intervention completion | up to 6 months (following 3 month timepoint collection for all subjects)
  RE-AIM interview guides will tailored to subjects, health coaches, and site personnel will solicit qualitative information for process evaluation, which is the primary purpose of this study.

SECONDARY OUTCOMES:
Change in patient activation | Baseline and 3 months
  The Patient Activation Measure is a 13-item scale designed for this purpose.
Change in subject perception of interpersonal support | Baseline and 3 months
  The Interpersonal Support Evaluation List (ISEL-12) will be used for this purpose.
Change in body mass index | Baseline and 3 months
  BMI will be calculated using height measurement from baseline, and weight measurements at baseline and then again at 3 months.

OTHER OUTCOMES:
Subject perception of community health-related resources and needs following intervention completion | up to 6 months (following 3 month timepoint for all subjects at the CAARE Inc. site))
  A focus group will provide qualitative data on subject perception of community resources and community health-related needs for those participants at the CAARE site who received health coaching.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Wolever, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Healing with CAARE Inc., Durham, North Carolina
  - Duke Healthy Lifestyles Program at Duke Children's Primary Care, Durham, North Carolina

REFERENCES:
- [Background] Seligman ME, Steen TA, Park N, Peterson C. Positive psychology progress: empirical validation of interventions. Am Psychol. 2005 Jul-Aug;60(5):410-21. doi: 10.1037/0003-066X.60.5.410. PMID 16045394
- [Background] Wolever RQ, Dreusicke M, Fikkan J, Hawkins TV, Yeung S, Wakefield J, Duda L, Flowers P, Cook C, Skinner E. Integrative health coaching for patients with type 2 diabetes: a randomized clinical trial. Diabetes Educ. 2010 Jul-Aug;36(4):629-39. doi: 10.1177/0145721710371523. Epub 2010 Jun 9. PMID 20534872
- [Background] Edelman D, Oddone EZ, Liebowitz RS, Yancy WS Jr, Olsen MK, Jeffreys AS, Moon SD, Harris AC, Smith LL, Quillian-Wolever RE, Gaudet TW. A multidimensional integrative medicine intervention to improve cardiovascular risk. J Gen Intern Med. 2006 Jul;21(7):728-34. doi: 10.1111/j.1525-1497.2006.00495.x. PMID 16808774
- [Background] Vorderstrasse AA, Ginsburg GS, Kraus WE, Maldonado MC, Wolever RQ. Health coaching and genomics-potential avenues to elicit behavior change in those at risk for chronic disease: protocol for personalized medicine effectiveness study in air force primary care. Glob Adv Health Med. 2013 May;2(3):26-38. doi: 10.7453/gahmj.2013.035. PMID 24416670
- [Background] Taggart J, Williams A, Dennis S, Newall A, Shortus T, Zwar N, Denney-Wilson E, Harris MF. A systematic review of interventions in primary care to improve health literacy for chronic disease behavioral risk factors. BMC Fam Pract. 2012 Jun 1;13:49. doi: 10.1186/1471-2296-13-49. PMID 22656188
- [Background] Holland SK, Greenberg J, Tidwell L, Malone J, Mullan J, Newcomer R. Community-based health coaching, exercise, and health service utilization. J Aging Health. 2005 Dec;17(6):697-716. doi: 10.1177/0898264305277959. PMID 16377768
- [Background] Holland SK, Greenberg J, Tidwell L, Newcomer R. Preventing disability through community-based health coaching. J Am Geriatr Soc. 2003 Feb;51(2):265-9. doi: 10.1046/j.1532-5415.2003.51068.x. PMID 12558726
- [Background] Steventon A, Tunkel S, Blunt I, Bardsley M. Effect of telephone health coaching (Birmingham OwnHealth) on hospital use and associated costs: cohort study with matched controls. BMJ. 2013 Aug 6;347:f4585. doi: 10.1136/bmj.f4585. PMID 23920348
- [Background] Rubin DL, Freimuth VS, Johnson SD, Kaley T, Parmer J. Training meals on wheels volunteers as health literacy coaches for older adults. Health Promot Pract. 2014 May;15(3):448-54. doi: 10.1177/1524839913494786. Epub 2013 Jul 22. PMID 23877229
- [Background] Nishita C, Cardazone G, Uehara DL, Tom T. Empowered diabetes management: life coaching and pharmacist counseling for employed adults with diabetes. Health Educ Behav. 2013 Oct;40(5):581-91. doi: 10.1177/1090198112465088. Epub 2012 Nov 21. PMID 23174629